CLINICAL TRIAL: NCT05344079
Title: Comparison of Epidural Analgesia and Local Infiltrative Analgesia
Brief Title: Comparison of the Effects of Epidural Analgesia and Local Infiltrative Analgesia Methods on Pain Control
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samsun Education and Research Hospital (Other)
Responsible Party: Principal Investigator, Hale Kefeli Celik, Anesthesiologist, Principal Investigator, Samsun Education and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KAEK-16/03-LIA
Record Dates: First submitted 2022-04-18; First posted 2022-04-25 (Actual); Last update posted 2022-04-29 (Actual); Status verified 2022-04

CONDITIONS: Epidural Anesthesia
Keywords: analgesia; knee arthroplasty; epidural; infiltrative; stress
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Epidural (Active Comparator): Patients in this group were entered the epidural space from the midline using the loss of resistance method with an 18-Gauge Touhy (Egemen®, Combifix Standard Spinal Epidural Combined Set, İzmir, Turkey) needle from the L4-L5 or L5-S1 vertebral space.
  Interventions: Device: 18-Gauge Touhy (Egemen®, Combifix Standard Spinal Epidural Combined Set, İzmir, Turkey)
- local infiltrative analgesia (Active Comparator): At the end of the operation, a 20-gauge infiltrative analgesia catheter connected to an ON-Q elastomeric pump that provides 5 mL/hour infusion prepared with 60 mL of 0.9% NaCl + 60 mL of 0.5% Bupivacaine (Bustesin®, 0.5% Spinal Heavy Vem Pharmaceuticals, Turkey) was placed on the fascia by the surgeon in such a way that all the holes of the catheter were under the skin and parallel to the incision line.
  Interventions: Device: 20-gauge infiltrative analgesia catheter connected to an ON-Q elastomeric pump

INTERVENTIONS:
Device: 18-Gauge Touhy (Egemen®, Combifix Standard Spinal Epidural Combined Set, İzmir, Turkey) — Patients in this group were entered the epidural space from the midline using the loss of resistance method with an 18-Gauge Touhy (Egemen®, Combifix Standard Spinal Epidural Combined Set, İzmir, Turkey) needle from the L4-L5 or L5-S1 vertebral space. After the free cerebrospinal fluid flow is observed by passing the spinal needle through the epidural needle, spinal anaesthesia was maintained with 10-15 mg hyperbaric bupivacaine (Bustesin®, 0.5% Spinal Heavy Vem Pharmaceuticals, Turkey). After the epidural catheter was fixed in such a way that it remained 5 cm in the epidural space, the adapter was inserted and fixed. Whether the catheter is in place or not was checked by 2 mL (40 mg) Lidocaine (Aritmal®, 2% 100 mg/5 mL amp., Biosel, Turkey) + 1/2000000 adrenaline test dose.
  Arms: Epidural
Device: 20-gauge infiltrative analgesia catheter connected to an ON-Q elastomeric pump — spinal anesthesia was maintained with 10-15 mg of hyperbaric bupivacaine (Bustesin 0.5% Spinal Heavy; Vem Pharmaceutical Industry and Trade Ltd.) after free cerebrospinal fluid flow was observed by entering the subarachnoid space with a 22 G spinal needle (Egemen Quincke Sharpened Spinal Anesthesia Needle; İzmir) from the L4-L5 or L5-S1 vertebral space. At the end of the operation, a 20-gauge infiltrative analgesia catheter connected to an ON-Q elastomeric pump that provides 5 mL/hour infusion prepared with 60 mL of 0.9% NaCl + 60 mL of 0.5% Bupivacaine (Marcaine 0.5%; AstraZeneca Industry and Trade Ltd.) was placed on the fascia by the surgeon in such a way that all the holes of the catheter were under the skin and parallel to the incision line. Pain pump and the catheter was withdrawn at the end of the postoperative 24th hour.
  Arms: local infiltrative analgesia

SUMMARY:
Total knee arthroplasty (TKA) is one of the major orthopedic surgeries that cause severe postoperative pain. 60% of the patients undergoing TKA have severe pain and 30% have moderate pain postoperatively. Many methods are used in the effective treatment of pain after TKA. The administration of analgesic drugs to the wound site in the form of local infiltration is included in the pain treatment both as an independent technique and in addition to multimodal analgesia in the treatment of postoperative pain. Epidural analgesia (EA) is known for its place in the treatment of pain after TKA and its suppressive effect on the stress response. Similar to the study, no publication was found in the literature that evaluated the suppression of surgical stress response and the effectiveness of local infiltrative analgesia (LIA) in lower extremity surgery. Therefore, it was aimed in the study to compare the effects of EA and LIA on postoperative pain and stress response in patients who underwent total knee arthroplasty.

DETAILED DESCRIPTION:
The study was planned as a prospective, randomized and single-center study, and the study was started after the approval of the local ethics committee. Informed consent form was obtained from each participants. All surgeries were performed before 11 am to ensure that the measurements of endocrine parameters matched the diurnal rhythm.

A total of 51 ASA I-III participants scheduled for TKA were randomly divided into two groups using the closed envelope method. Groups were group E administered epidural analgesia (n=25) and group I local infiltrative analgesia (n=26). After an overnight fasting period, the participants who were taken to the operating room were hydrated with 500 mL of saline 30 minutes before the operation, and no premedication was applied to the patients. When the participants were taken to the operating table, routine ECG (DII), non-invasive blood pressure, and peripheral oxygen saturation were monitored.

The same surgical technique was performed by the same surgeon in both groups. The same prosthesis was used in both groups, 750 mg cefuroxime iv. for prophylactic antibiotics (Cefax; Vem Pharmaceutical Industry and Trade Ltd.) and the patients were administered diclofenac sodium 75 mg regularly every 12 hours (Diclomec; Abdi İbrahim Pharmaceuticals Ind. and Trade Inc.).

Group E: Participants in this group were entered the epidural space from the midline using the loss of resistance method with an 18-Gauge Touhy (Egemen Combifix Standard Spinal Epidural Combined Set; Braun) needle from the L4-L5 or L5-S1 vertebral space. After the free cerebrospinal fluid flow is observed by passing the spinal needle through the epidural needle, spinal anaesthesia was maintained with 10-15 mg hyperbaric bupivacaine (Bustesin 0.5% Spinal Heavy; Vem Pharmaceuticals Industry and Trade Ltd.). After the epidural catheter was fixed in such a way that it remained 5 cm in the epidural space, the adapter was inserted and fixed. Whether the catheter is in place or not was checked by 2 mL (40 mg) Lidocaine (Aritmal; Osel Pharmaceuticals Ind. Inc.) + 1/2000000 adrenaline test dose. At the end of the surgery, when the Bromage score is 2 in the recovery room, 60 mL 0.9% NaCl + 0.5% 60 mL bupivacaine (Marcaine 0.5%; AstraZeneca Industry and Trade Ltd.) was inserted into the epidural catheter to provide continuous infusion at a rate of 5 mL/hour, and the participants were followed in the postanesthetic care unit for 24 hours.

Group I: In this group, spinal anesthesia was maintained with 10-15 mg of hyperbaric bupivacaine (Bustesin 0.5% Spinal Heavy; Vem Pharmaceutical Industry and Trade Ltd.) after free cerebrospinal fluid flow was observed by entering the subarachnoid space with a 22 G spinal needle (Egemen Quincke Sharpened Spinal Anesthesia Needle; İzmir) from the L4-L5 or L5-S1 vertebral space. At the end of the operation, a 20-gauge infiltrative analgesia catheter connected to an ON-Q elastomeric pump that provides 5 mL/hour infusion prepared with 60 mL of 0.9% NaCl + 60 mL of 0.5% Bupivacaine (Marcaine 0.5%; AstraZeneca Industry and Trade Ltd.) was placed on the fascia by the surgeon in such a way that all the holes of the catheter were under the skin and parallel to the incision line. When the Bromage score was 2 in the postoperative recovery room, drug infusion was started with an incisional pain pump and the catheter was withdrawn at the end of the postoperative 24th hour.

Bromage score used in participants in the epidural analgesia group; 0: No paralysis, the patient can move his foot and knee fully; 1: The patient only moves his knee and foot, cannot raise his leg straight; 2: The patient cannot move the knee, only the ankle; 3: It was evaluated as complete paralysis.

In the postoperative period in participants 4th, 6th, 12th, pain at rest and with movement (passive flexion movement to the knee joint at the operation site) was measured with the Visual Analog Scale (VAS) at the 24th. VAS assessment was done by asking the participants to mark a point on a 10 cm horizontal line that shows (initial "no pain", end "unbearable pain") the start and end points and is equivalent to the pain on this line. In both groups, if the VAS value is 4 and above, 50 mg iv. tramadol hydrochloride (Contromal; Abdi İbrahim Pharmaceuticals Ind. and Trade Inc.) additional dose was administered.

Tramadol hydrochloride consumption and side effects were evaluated as nausea (0=absent, 1=mild, 2=severe) and vomiting (0=absent, 1=mild, 2=severe). The presence of urinary retention and abdominal distension was recorded. Venous blood samples were taken in the preoperative period, at the 1st hour, 4th hour, and 24th hour postoperatively to evaluate the stress response.

ELIGIBILITY:
Inclusion Criteria: Patients,

* ASA II and III,
* Aged between 18-80 years,
* who were scheduled to undergo unilateral knee arthroplasty,
* who giving consent.

Exclusion Criteria: Patients

* who will undergo an extra surgical procedure or who will undergo bilateral knee arthroplasty,
* those with local anaesthetic sensitivity,
* morbidly obese,
* those with additional pathology that may constitute a contraindication to the application of regional anaesthesia,
* those who did not give voluntary consent,
* had a history of anticoagulant drug use,
* had a history of cerebrovascular disease,
* who received steroid therapy for any disease, were diabetic,
* had a homeostasis assessment score (HOMA) above 2.5.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — It is known that gender difference is different in both stress response and pain perception. Therefore, only female patients and patients who will undergo a single TKA were included in the study in order to standardize the study. (Rosen S, Ham B, Mogil JS. Sex differences in neuroimmunity and pain. J Neurosci Res 2017;95:500-508)
Enrollment: 51 (Actual)
Dates: Start 2016-05-01 (Actual); Primary Completion 2017-03-03 (Actual); Study Completion 2017-05-01 (Actual)

PRIMARY OUTCOMES:
Visual analog scale | From 4 hours to 24 hours postoperative
  Following surgery, the patient's pain level will be recorded in a visual analog scale (VAS) at 4 hours, 6 hours, 12 hours, 24 hours. VAS assessment was done by asking the patient to mark a point on a 10 cm horizontal line that shows (initial "no pain", end "unbearable pain") the start and end points and is equivalent to the pain on this line.

CONTACTS AND LOCATIONS:
Overall Officials: Zahide Doganay, Professor, Study Chair — Samsun Research and Education Hospital
Locations (1):
- Samsun Research and Education Hospital, Samsun, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Researched data and statistical analyzes will be available from the journal in which the clinical study was published.

REFERENCES:
- [Result] Berninger MT, Friederichs J, Leidinger W, Augat P, Buhren V, Fulghum C, Reng W. Effect of local infiltration analgesia, peripheral nerve blocks, general and spinal anesthesia on early functional recovery and pain control in total knee arthroplasty. BMC Musculoskelet Disord. 2018 Jul 18;19(1):232. doi: 10.1186/s12891-018-2154-z. PMID 30021587
- [Result] Peng XQ, Fei ZG, Sun CG, Zhou QJ. Efficacy and safety of local infiltration analgesia for pain management in total knee and hip arthroplasty: A meta-analysis of randomized controlled trial. Medicine (Baltimore). 2020 May 29;99(22):e20640. doi: 10.1097/MD.0000000000020640. PMID 32481477
- [Result] Gibbison B, Angelini GD, Lightman SL. Dynamic output and control of the hypothalamic-pituitary-adrenal axis in critical illness and major surgery. Br J Anaesth. 2013 Sep;111(3):347-60. doi: 10.1093/bja/aet077. Epub 2013 May 9. PMID 23661405
- [Result] Fusco P, Cofini V, Petrucci E, Scimia P, Fiorenzi M, Paladini G, Behr AU, Borghi B, Flamini S, Pizzoferrato R, Colafarina O, Di Francesco A, Tabacco T, Necozione S, Marinangeli F. Continuous wound infusion and local infiltration analgesia for postoperative pain and rehabilitation after total hip arthroplasty. Minerva Anestesiol. 2018 May;84(5):556-564. doi: 10.23736/S0375-9393.17.12110-3. Epub 2017 Oct 4. PMID 28984095
- [Result] Li C, Qu J, Pan S, Qu Y. Local infiltration anesthesia versus epidural analgesia for postoperative pain control in total knee arthroplasty: a systematic review and meta-analysis. J Orthop Surg Res. 2018 May 16;13(1):112. doi: 10.1186/s13018-018-0770-9. PMID 29769140